CLINICAL TRIAL: NCT01275001
Title: Effects of Music Intervention on the Brain Development of Preschool Children
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AIHBG-1360-MRI
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-01

CONDITIONS: Child Development
Keywords: brain; brain development; MRI; preschool children; cortical mantle thickness; hippocampal volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention children: Children who are receiving a Suzuki-like violin instruction through their participation in an Early Childhood/Headstart preschool program
- Control Group: Preschool-age children who are not receiving Suzuki-like violin instruction

SUMMARY:
The purpose of this research study is to learn more about the effects a musical intervention has on typical brain development in preschool-aged children.

DETAILED DESCRIPTION:
This study will advance the science on brain research in young children by determining the effects of a musical intervention or training on children's brain development. The study will investigate how regular instruction in the Suzuki-like method of violin affects brain structure and function over the course of approximately five (5) months in preschool-aged children participating in an Early Childhood/Headstart preschool program when compared to a control group of their peers.

ELIGIBILITY:
Inclusion Criteria:

* Children who are between the ages of 3 and 4.5 years old and are involved in the intervention arm of the Avera Family Wellness Program
* Children who are between the ages of 3 and 4.5 years old and are involved in the control arm of the Avera Family Wellness Program

Exclusion Criteria:

* Unable to provide written consent to participate in the research project
* Unable to complete the MRI scan

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants in this research project will be involved with a different research project (Avera Family Wellness Program) investigating the effects of a family-based wellness approach to addressing emotional-behavioral needs of preschool-age children and their families. The Avera Family Wellness Program (AFWP) consists of a group of children who receive the family-based intervention and a group of control preschool-age children.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cortical mantle thickness | 5 months
  Measure cortical mantle thickness in unsedated preschool-age children with an initial magnetic resonance imaging (MRI) scan and compare to measured cortical mantle thickness after a second MRI scan in the same children after 5 months

SECONDARY OUTCOMES:
Hippocampal volume | 5 months
  Measure hippocampal volumes in unsedated preschool-age children with an initial MRI scan and compare hippocampal volumes in the same children with a second MRI scan after 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Soundy, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Ho YC, Cheung MC, Chan AS. Music training improves verbal but not visual memory: cross-sectional and longitudinal explorations in children. Neuropsychology. 2003 Jul;17(3):439-50. doi: 10.1037/0894-4105.17.3.439. PMID 12959510
- [Background] Samson S, Peretz I. Effects of prior exposure on music liking and recognition in patients with temporal lobe lesions. Ann N Y Acad Sci. 2005 Dec;1060:419-28. doi: 10.1196/annals.1360.035. PMID 16597796
- [Background] Fujioka T, Ross B, Kakigi R, Pantev C, Trainor LJ. One year of musical training affects development of auditory cortical-evoked fields in young children. Brain. 2006 Oct;129(Pt 10):2593-608. doi: 10.1093/brain/awl247. Epub 2006 Sep 7. PMID 16959812
- [Background] Peterson BS. Neuroimaging in child and adolescent neuropsychiatric disorders. J Am Acad Child Adolesc Psychiatry. 1995 Dec;34(12):1560-76. doi: 10.1097/00004583-199512000-00006. PMID 8543527
- [Background] Durston S, Tottenham NT, Thomas KM, Davidson MC, Eigsti IM, Yang Y, Ulug AM, Casey BJ. Differential patterns of striatal activation in young children with and without ADHD. Biol Psychiatry. 2003 May 15;53(10):871-8. doi: 10.1016/s0006-3223(02)01904-2. PMID 12742674
- [Background] Symms M, Jager HR, Schmierer K, Yousry TA. A review of structural magnetic resonance neuroimaging. J Neurol Neurosurg Psychiatry. 2004 Sep;75(9):1235-44. doi: 10.1136/jnnp.2003.032714. PMID 15314108
- [Background] Gogtay N, Giedd JN, Lusk L, Hayashi KM, Greenstein D, Vaituzis AC, Nugent TF 3rd, Herman DH, Clasen LS, Toga AW, Rapoport JL, Thompson PM. Dynamic mapping of human cortical development during childhood through early adulthood. Proc Natl Acad Sci U S A. 2004 May 25;101(21):8174-9. doi: 10.1073/pnas.0402680101. Epub 2004 May 17. PMID 15148381